CLINICAL TRIAL: NCT06562309
Title: Fecal Microbiota and Monocyte Trained Immunity in Patients With Coronary Heart Disease and Different Level of High-sensitivity C-reactive Protein (hsCRP)
Brief Title: Fecal Microbiota and Monocyte Trained Immunity in CHD Patients With Different hsCRP
Status: Completed | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiang Cheng, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: Trainedmono
Record Dates: First submitted 2024-08-14; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Coronary Heart Disease; Unstable Angina
MeSH Terms: conditions — Coronary Disease; Angina, Unstable

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high inflammatory risk: hsCRP ≥ 3mg/L
  Interventions: Other: take feces and blood samples from patients
- low inflammatory risk: hsCRP < 1mg/L
  Interventions: Other: take feces and blood samples from patients

INTERVENTIONS:
Other: take feces and blood samples from patients — this study does not involve any intervention

SUMMARY:
This single-center study enrolled patients aged 35-75 years who were diagnosed with unstable angina (UA), and had at least one of the three major coronary arteries with a ≥ 50% reduction in lumen diameter by angiographic visual estimation. Patients were all recruited at the Department of Cardiology, Union Hospital, Wuhan, Hubei Province, China. Feces and blood samples were collected on admission were used promptly for ex vivo studies.

DETAILED DESCRIPTION:
This single-center study enrolled patients aged 35-75 years who were diagnosed with unstable angina (UA), and had at least one of the three major coronary arteries with a ≥ 50% reduction in lumen diameter by angiographic visual estimation. Patients were all recruited at the Department of Cardiology, Union Hospital, Wuhan, Hubei Province, China. Exclusion criteria included acute myocardial infarction, prior myocardial infarction, malignancies, auto-immune or auto-inflammatory diseases, or ongoing infection. Feces and blood samples were collected on admission were used promptly for ex vivo studies.

the aim of the study is to investigate whether the fecal microbiota and peripheral blood monocytes in patients with coronary heart disease at different levels of inflammation are associated with the level of inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Age >35 and <75 years
2. Admitted for UA and had at least one of the three major coronary arteries with ≥50% reduction in lumen diameter by angiographic visual estimation
3. Informed consent obtained

Exclusion Criteria:

1. Prior myocardial infarction
2. Left ventricular ejection fraction ≤ 40% on echocardiography
3. Have a history of malignancies, auto-immune, auto-inflammatory disease or on immunomodulatory medication
4. Ongoing acute, chronic, or concurrent infectious disease
5. Surgery 3 months before sample collection
6. Immunization with a vaccine within 4 weeks before sample collection
7. Pregnancy, or breast feeding
8. History of primary or secondary immunodeficiency
9. Renal failure with estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m2
10. Active liver disease with alanine aminotransferase (ALT >80 U/L) or aspartate aminotransferase (AST > 80 U/L)
11. History of chronic obstructive pulmonary disease (COPD)
12. Refuse to provide written consent
13. Any other circumstances in which the investigator judges that the patient is not suitable

Ages: 35 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants This single-center study enrolled patients aged 35-75 years who were diagnosed with UA, and had at least one of the three major coronary arteries with a ≥ 50% reduction in lumen diameter by angiographic visual estimation. Patients were all recruited at the Department of Cardiology, Union Hospital, Wuhan, Hubei Province, China. UA diagnosis followed the 2014 AHA/ACC Guideline.18 Exclusion criteria included acute myocardial infarction, prior myocardial infarction, malignancies, auto-immune or auto-inflammatory diseases, or ongoing infection. Feces and blood samples were collected on admission were used promptly for ex vivo studies.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
blood monocytes trained immunity | within 3 days
  1.Blood monocytes were detected by flowcytometry to evaluate the monocyte subsets and CCR2 expression; 2. monocytes were enriched from blood cells and used for ex vivo lipopolysaccharide stimulation, mRNA sequencing and ATAC sequencing; 3.The metabolic bias of monocytes was detected by Seahorse technology and metabolics.

SECONDARY OUTCOMES:
fecal microbiome profile | within 3 days
  the feccal microbiota was detected by 16s rRNA sequencing, and the analyses includes alpha and beta diversity, the differential microbiota between two groups, and the correlation between microbiota and clinical characteristics including age, BMI, blood lipids, and other available continous variables.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Cheng, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
The data and material are accessible in proper request.